CLINICAL TRIAL: NCT00306397
Title: Open, Single Centre, Pilot Study to Investigate a Steroid Free Immunosuppressive Regimen for De Novo Renal Transplant Recipients Followed by Randomisation to Calcineurin Inhibitor Containing or Calcineurin Inhibitor Free Immunosuppression
Brief Title: Pilot Study to Investigate a Steroid Free Immunosuppressive Regimen for Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Steiger Juerg / Professor, University Hospital Basel, Clinic for transplantation immunology and nephrology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL-080-CH02; 2004DR3379
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Steroid free; Calcineurin inhibitor free; Tacrolimus; Sirolimus
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Rapamycin - MMF after 3 months
  Interventions: Drug: Rapamycin
- B (Active Comparator): Low dose tacrolimus - MMF - Rapamycin after 3 months
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Sirolimus perorally following kidney transplantation, randomisation after protocol biopsy at months three to a) Sirolimus - MF- or b) low dose tacrolimus - sirolimus -MMF -
  Other Names: Sirolimus; Rapammune

SUMMARY:
The main purpose of this study is to investigate, whether a steroid free immunosuppressive treatment is a valuable alternative in the treatment of de novo kidney transplant recipients and if it is possible to withdraw calcineurin inhibitors after 3 months.

DETAILED DESCRIPTION:
Protocol synopsis Title An open, single centre, pilot study to investigate a steroid free immunosuppressive regimen for de novo renal transplant recipients followed by a two arm randomization to a calcineurin inhibitor containing and a calcineurin inhibitor free maintenance immunosuppression after three months. Study code Sterfree pilot study Project phase An open, single centre, one arm study followed by a 1:1 randomized, parallel group, comparative study after three months. Study objectives To obtain preliminary information on the efficacy and safety of a rapamycin / sodium-mycophenolate (Myfortic) / tacrolimus regimen in the absence of steroids for the prevention of acute rejection following renal transplantation. To compare a low dose tacrolimus / rapamycin / sodium-mycophenolate (Myfortic) regimen to a rapamycin / sodium-mycophenolate regimen in patients without evidence of acute rejection after three months.

Efficacy:

Primary endpoint

* Plasma creatinine (and creatinine clearance (Cockcroft)) Secondary endpoints
* Incidence of first acute rejections and total number of acute rejections
* Total number of anti-rejection treatments
* Patients successfully withdrawn from calcineurin inhibitor at three months
* Graft survival
* Patient survival

Safety:

* Graft survival
* Patient survival
* Protocol biopsies at 3 months( range: day 75 to 105) and 6 months (range day 165 to 195) sub clinical rejection
* Incidence of first acute biopsy proven rejection and total number of acute rejection episodes
* Total number of anti-rejection treatments
* Patients switched from assigned therapy due to rejection or side effects
* Patients needing steroids because of rejection
* Incidence of selected adverse events: tubulointerstitial nephrotoxicity (TOR inhibitor), leucopenia, thrombocytopenia, elevated fasting blood glucose, dyslipidemia, , electrolyte disturbances, de novo insulin dependency, gastrointestinal disorders (non infectious), neurotoxicity.
* Patients withdrawn due to adverse events

Long term patient follow up Patients will be followed up for graft and patient survival at 12, 24, and 36 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with end stage kidney disease suitable for primary renal transplantation or retransplantation
* patients receiving a graft from a living related, living unrelated or brain-death donor

Exclusion Criteria:

* patients with a low or high immunological risk constellation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Allograft function | 6 months

SECONDARY OUTCOMES:
Patients successfully withdrawn from calcineurin inhibitor after three months | 3 months
Graft survival | 6 months
Patient survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Juerg U Steiger, MD, Principal Investigator — University Hospital Basel, Clinic for Transplantation Immunology and Nephrology
Locations (1):
- University Hospital Basel, Clinic for Transplantation Immunology and Nephrology, Basel, Switzerland